CLINICAL TRIAL: NCT00972790
Title: Effect of Bilateral Scalp Nerve Blocks on Post-operative Pain and Discharge Times in Patients Undergoing Supra-tentorial Craniotomy and General Anaesthesia
Brief Title: Scalp Nerve Blocks for Post-Craniotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-0041-GAP
Record Dates: First submitted 2009-09-04; First posted 2009-09-09 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2011-12

CONDITIONS: Supratentorial Neoplasms; Aneurysms; Arteriovenous Malformation; Epilepsy
Keywords: brain tumor; un-ruptured aneurysm; arteriovenous malformation; epileptic focus; supratentorial
MeSH Terms: conditions — Supratentorial Neoplasms; Aneurysm; Arteriovenous Malformations; Epilepsy; Brain Neoplasms | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Sham Comparator): The patients in the control arm will receive sham nerve blocks with 20 ml of saline + epinephrine 1:200,000, in a manner identical to that described for the treatment group.
  Interventions: Procedure: Bilateral Scalp Nerve Blocks
- Intervention Group (Active Comparator): The patients in the intervention group will receive bilateral scalp nerve blocks with a total of 20 ml of 0.5% bupivacaine + epinephrine 1:200,000.
  Interventions: Procedure: Bilateral Scalp Nerve Blocks

INTERVENTIONS:
Procedure: Bilateral Scalp Nerve Blocks — Scalp nerve blocks will be performed bilaterally at the end of the surgery under general anaesthesia and before removal of the head holder. Patients will receive scalp nerve blocks with a total of 20 ml of 0.5% bupivacaine + epinephrine 1:200,000 or 20 ml of saline + epinephrine 1:200,000. Solution volume is as follows: 2ml each bilaterally for supraorbital and supratrochlear nerves; 3 ml for the auriculotemporal nerves; 2 ml for the postauricular branches of the greater auricular nerves and for the greater, lesser, and third occipital nerves 3 ml of solution will be infiltrated along the superior nuchal line, approximately halfway between the occipital protuberance and the mastoid process.
  Other Names: 0.5% Marcaine; Normal Saline

SUMMARY:
The objective of this study is to demonstrate that scalp nerve blocks ("scalp freezing"), performed at the end of supratentorial brain surgery, will reduce post-operative pain, opioids side effects, and the time required for post-anaesthesia care unit (PACU)/Intensive Care Unit (ICU) and hospital discharge.

DETAILED DESCRIPTION:
The proposed study is a randomized, placebo-controlled, triple-blinded, parallel-group clinical trial. Patients will be recruited from the neurosurgical population at St. Michael's Hospital.

The inclusion criteria are:

* Adults aged 18 years and over;
* scheduled for one of the following supratentorial craniotomy:

  1. resection of a brain tumour
  2. clipping of an un-ruptured cerebral aneurysm
  3. excision of an artero-venous malformation (AVM), or
  4. removal of an epileptic focus
* ASA physical status < IV

Intervention group: scalp nerve blocks with 20 ml of bupivacaine 0.5% + epinephrine 1:200,000 (divided among the different injection sites) at the end of surgery and before removal of the endo-tracheal tube. Control group: equal injections with 20 ml of saline + epinephrine 1:200,000 (at same time). In both study arms, post-operative rescue analgesia will be provided with hydromorphone patient-controlled analgesia (PCA).

The primary outcome of this study will be the 24h post-operative pain score as assessed by the visual analogue scale (VAS).

Important secondary outcomes will be:

* the total PCA hydromorphone consumption in the first 24 and 48 post-operative hours;
* the incidence of nausea and vomiting in the first 24 and 48 post-operative hours;
* time to reach discharge eligibility from the PACU/ICU and hospital length of stay.

Patients will be asked to rate their pain using the VAS at 30 min, 1, 2, 4, 8, 12, 18, 24, and 48 h, postoperatively by the research coordinator/bedside nurse. Pain will be also assessed at 5, 30 and 60 days postoperatively with the use of a Numeric Rating Scale (0-10).

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years and over;
* patients scheduled for elective craniotomy under general anaesthesia for one of the following surgeries:

  * resection of a supratentorial brain tumour,
  * clipping of an un-ruptured supratentorial cerebral aneurysm,
  * excision of a supratentorial arterio-venous malformation (AVM),
  * removal of an epileptic focus under general anaesthetic.
* ASA physical status < IV.

Exclusion Criteria:

* history of significant coronary artery disease (NYHA class III or IV) which would contraindicate the use of epinephrine;
* presence of pain related to the intracranial pathology (e.g. tumour pain) since it could make difficult the discrimination between the tumour pain itself and the surgery related pain;
* current history of alcohol abuse or recreational drug abuse;
* active psychotic disorder;
* history of chronic pain requiring chronic opioids use (patients on opioids for > 2 weeks);
* known or suspected addiction to narcotic substances;
* presence of any acute distracting pain;
* history of migraines;
* inability to understand or incapacity to use the VAS;
* proven or suspected allergy to local anaesthetics;
* craniotomy incision extending beyond the field of the block;
* predicted need for postoperative ventilation;
* history of scalp paresthesia or scalp scarring that may preclude normal nerve anatomy;
* previous craniotomy or cranial irradiation;
* history of malignant hyperthermia, which would contraindicate the anaesthesia maintenance protocol of this study;
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the 24h post-operative VAS score among adults undergoing supratentorial craniotomy. | 24 hours

SECONDARY OUTCOMES:
48h post-operative pooled VAS score | 48 hours
the total PCA hydromorphone consumption in the first at 24 and 48 post-operative hours | 24 and 48 hours
total hydromorphone demands and delivered doses in the first 24 and 48 post-operative hours | 24 and 48 hours
the incidence of nausea and vomiting in the first 24 and 48 post-operative hours | 24 and 48 hours
the time for patients to reach discharge eligibility from the PACU/ICU | Discharge time and date from PACU/ICU
the time for patients to reach discharge eligibility from hospital | Discharge time and date from hospital
presence of long term pain as measured with the Numeric Rating Scale (NRS) at days 5, 30 and 60 postoperatively | 5, 30 and 60 days
Karnofsky Performance Scale Index and modified pain treatment satisfaction scale (PTSS) at day 5 | day 5

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Rigamonti, MD, MSc (c), Principal Investigator — St. Michael's Hospital, University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Rigamonti A, Garavaglia MM, Ma K, Crescini C, Mistry N, Thorpe K, Cusimano MD, Das S, Hare GMT, Mazer CD. Effect of bilateral scalp nerve blocks on postoperative pain and discharge times in patients undergoing supratentorial craniotomy and general anesthesia: a randomized-controlled trial. Can J Anaesth. 2020 Apr;67(4):452-461. doi: 10.1007/s12630-019-01558-7. Epub 2019 Dec 26. PMID 31879855